CLINICAL TRIAL: NCT05754450
Title: A Phase 3, Open-Label, Extension Study to Assess the Long-term Safety and Efficacy of AVTX-803 in Subjects with Leukocyte Adhesion Deficiency Type II (LAD II)
Brief Title: An Extension Study Assessing the Safety and Efficacy of AVTX-803 in Subjects with Leukocyte Adhesion Deficiency Type II
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AUG Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AVTX-803-LAD-302
Record Dates: First submitted 2023-02-06; First posted 2023-03-03 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-03

CONDITIONS: Leukocyte Adhesion Deficiency
MeSH Terms: conditions — Leukocyte adhesion deficiency type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- AVTX-803 (Experimental): AVTX-803 at a dose specified by the investigator up to 5 times a day not to exceed 1700 mg/kg/day
  Interventions: Drug: AVTX-803

INTERVENTIONS:
Drug: AVTX-803 — L-fucose crystalline powder

SUMMARY:
The primary objective of this extension study is to assess the long-term safety and efficacy of AVTX-803 in subjects with LAD II (SLC35C1-CDG).

ELIGIBILITY:
Inclusion Criteria:

* Subject must have completed protocol AVTX-803-LAD-301
* Subject has biochemically and genetically proven LAD II (SLC35C1-CDG)

Exclusion Criteria:

* Subject has severe anemia defined as hemoglobin <8.0 g/dL (<4.9 mmol/L)
* Subject has impaired renal function as defined by an eGFR <90 mL/min
* Subject has known or suspected intolerance or hypersensitivity to fucose or any ingredients of the investigational product
* In the investigator's opinion, subject has a history of failure to respond to fucose at adequate dosing

Ages: 6 Months to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Estimated)
Dates: Start 2023-04-10 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment emergent adverse events reported during the study attributable to AVTX-803. | Through study completion, an average of 1 year.

SECONDARY OUTCOMES:
Sialyl-Lewis X antigen expression on leukocytes | At 6 months
Change from Baseline in the composite Nijmegen Pediatric Congenital Disorders of Glycosylation (CDG) Rating Scale (NPCRS) | Through study completion, an average of 1 year.
  The NPCRS comprises 3 sections, with each section containing specific items relevant to the assessment of subjects with CDG. Section I (Current Function); Section II (System Specific Involvement); and Section III (Current Clinical Assessment). The sum of the scores is used to scale patients into 3 domains: mild (0-14), moderate (15-25), and severe (>26) category.
Change from Baseline in the individual parameters of the Nijmegen Pediatric Congenital Disorders of Glycosylation (CDG) Rating Scale (NPCRS) | Through study completion, an average of 1 year.
  The NPCRS comprises 3 sections, with each section containing specific items relevant to the assessment of subjects with CDG. Section I (Current Function); Section II (System Specific Involvement); and Section III (Current Clinical Assessment). The sum of the scores is used to scale patients into 3 domains: mild (0-14), moderate (15-25), and severe (>26) category.
Goal Attainment Score (GAS) | Through study completion, an average of 1 year.
  The parent (or subject) formulates 3 individual goals for improving quality of life. Typically, these goals affect mobility, independence, and disease-related health aspects. These goals will be re-evaluated and scored by the parent or subject at each study visit within a scale of -2 to +2.
Clinician Global Impression of Severity (CGI-S) | Through study completion, an average of 1 year.
  The CGI-S scale is a 7-point scale that assesses the severity of the subject's severity of disease/illness. 1=Normal, not ill at all; 2=borderline ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6= severely ill; 7=among the most extreme ill."

CONTACTS AND LOCATIONS:
Overall Officials: David Deyle, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No